CLINICAL TRIAL: NCT05147181
Title: Lanadelumab Treatment Outcomes in HAE Polish Patients Treated in the Scope of National Drug Program (NDP). Prospective, Multicenter Observational Study
Brief Title: A Study With Lanadelumab in Persons With Hereditary Angioedema (HAE) in Poland
Acronym: CHOPIN
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4003; MACS-2020-081003 (Other: Takeda)
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With HAE: Participants with type 1 or type 2 HAE when treated with lanadelumab in real life in accordance with Summary of Product Characteristics (SmPC) and NDP requirements will be observed in this prospective observational study for 36 months

SUMMARY:
The main aim of this study is to learn about how many persons with HAE type I or type II are attack-free when treated with lanadelumab in real life, how many attacks occur and how many of these attacks need rescue treatment and about the nature of HAE attacks.

Participants will need to visit their doctor 5 times in total as part of this study. The visits are planned every 6 months. Participants will also be asked to fill out questionnaires as part of this study.

ELIGIBILITY:
Inclusion Criteria

Participant eligibility is determined according to the following criteria prior to entry into the study:

* In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
* The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* HAE participant (aged greater than or equal to [>=] 12 years old.) qualified to treatment with lanadelumab in the NDP and receiving treatment according to the Summary of Product Characteristics for Takhzyro.
* Male or female participants, aged >=12 years old.

Exclusion Criteria

Any participant who meets any of the following criteria will not qualify for entry into the study:

* Currently participates or plans to participate in any interventional clinical trial.
* Any other reason that, in the Investigator's opinion, makes the participant unsuitable to participate in this study.

Participants should be included in the study only once. Data erroneously collected from participants for which written consent is not available, will not be included in or will be deleted from the database.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with HAE are included in this study.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Total Number of HAE Attacks to 3 Months on Lanadelumab Therapy | Baseline up to 3 months
  Change from baseline (3 months period prior to qualification to NDP) to 3 months on lanadelumab therapy in the total number of HAE attacks will be analyzed using either a Poisson or negative binomial mixed effect model with period (pre or post qualification to NDP) as fixed effect and participant as a random effect. Choice of modelling method will depend on the degree of overdispersion in number of HAE attacks.
Percentage of Participants Without HAE Attacks at Month 6 | At Month 6
  Percentage of participants without HAE attacks will be analyzed and reported at Month 6.
Percentage of Participants Without HAE Attacks at Month 12 | At Month 12
  Percentage of participants without HAE attacks will be analyzed and reported at Month 12.
Percentage of Participants Without HAE Attacks at Month 18 | At Month 18
  Percentage of participants without HAE attacks will be analyzed and reported at Month 18.
Percentage of Participants Without HAE Attacks at Month 24 | At Month 24
  Percentage of participants without HAE attacks will be analyzed and reported at Month 24.
Number of Participants Based on Type of Rescue Treatment Received | Up to 24 months
  Number of participants based on type of rescue treatment received will be analyzed and reported.
Percentage of Participants With HAE Attacks Who Received Rescue Treatment | Up to 24 months
  Percentage of participants with HAE attacks who received rescue treatment will be analyzed and reported.
Number of Participants Based on Severity of HAE Attacks | Up to 24 months
  Number of Participants based on severity of HAE Attacks i.e mild, moderate and severe will be analyzed. Mild means temporary or mild discomfort, moderate means activity limited mildly or moderately and some assistance may be needed and severe means activity considerably limited, assistance needed.
Number of Participants Based on Anatomical Location of HAE Attacks | Up to 24 months
  Number of participants based on anatomical location of HAE attacks per body part(s) affected, such as peripheral (e.g., skin), abdominal, upper airway (e.g., larynx), other organs, duration of symptoms/ number of days with angioedema symptoms will be analyzed and reported.
Time to First HAE Attack Requiring Rescue Treatment | Up to 24 months
  Kaplan-Meier analysis will be prepared for time to first HAE attack for which rescue treatment was used and time to first HAE attack after lanadelumab treatment discontinuation.
Percentage of Participants With HAE Attacks Based on Visit to Healthcare Professional (HCP), Electronic Record (ER) or Hospitalizations | Up to 24 months
  Percentage of participants with HAE Attacks will be analyzed and reported based on Visit to HCP, access to an ER or hospitalizations.
Duration of HAE Attack | Up to 24 months
  Duration of HAE Attack will be analyzed and reported.

SECONDARY OUTCOMES:
Number of Participants Categorized Based on Lanadelumab Treatments Patterns | Up to 24 months
  Number of participants categorized based on lanadelumab treatments patterns will be analyzed and reported.
Number of Participants Who Received Lanadelumab Treatment Prior to Discontinuation | Up to 24 months
  Number of participants who received lanadelumab treatment prior to discontinuation will be analyzed and reported.
Number of Participants Based on Reason for Lanadelumab Treatment Discontinuation | Up to 24 months
  Number of participants based on reason for lanadelumab treatment discontinuation will be analyzed and reported.
Change From Baseline in Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH) at End of Landelumab Therapy | Up to 24 months
  The WPAI:GH is a generic questionnaire to measure the effect of general health and symptom severity on work productivity and regular activities during the past seven days. It can be self or interviewer-administered to adults aged 18 years or older. This six-item PRO instrument covers work (five items) and daily activities (one item) using yes/no or numerical answers (number of hours). It takes approximately two to three minutes to complete. WPAI:GH outcomes are expressed as impairment percentages. An overall work productivity score (health or symptom) [%WP], is calculated by multiplying the percentage of work time spent working (health or symptom) [% WTW] by the percentage productivity at work (health or symptom) [%PW]: %WP = %WTW*%PW. High scores indicate prolonged sick leave or impairment and decreased productivity. Change from baseline to the end of lanadelumab therapy in WPAI:GH will be modelled with a linear model using baseline total score and time of therapy as predictors.
Change From Baseline in Angioedema Quality of Life (AE-QoL) at End of Landelumab Therapy | Up to 24 months
  Angioedema quality of life (AE-QoL) questionnaire was a self-administered validated angioedema disease-specific quality of life instrument. It consisted of 17 specific questions that were associated with work, physical activity, free time, social relations, and diet. Each of the 17 items had a 5-point response scale ranging from 1 (Never) to 5 (Very Often). The questionnaire was scored according to the developers' guidelines to produce a total score and 4 domain scores (functioning, fatigue/mood, fear/shame, nutrition). Raw domain scores (mean of the item scores within each scale) and the raw total score (mean of all item scores) were rescaled using linear transformations into final percentage scores ranging 0 to 100, based on the maximum possible score, where the higher the score the greater the QoL impairment. Change from baseline in AE-QOL at end of landelumab therapy will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- Poland (14):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeylandów/Szpital w Poznaniu, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki nr 2, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. Stefana Kardynała Wyszyńskiego, Lublin, Lublin Voivodeship
  - Wojskowy Instytut Medyczny, Warsaw, Masovian Voivodeship
  - Kliniczny Szpital Wojewódzki nr 1 im. Fryderyka Chopina w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok, Podlaskie Voivodeship
  - Uniwersytet Medyczny w Białymstoku, Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Zespół Gruźlicy i Chorób Płuc w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - SPSK nr 2 PUM w Szczecinie, Szczecin, Zachodniopomorske
  - SAMODZIELNY PUBLICZNY ZAKŁAD OPIEKI ZDROWOTNEJ - Centralny Szpital Kliniczny Uniwersytety Medycznego w Łodzi, Lodz, Łódź Voivodeship
  - Szpital Powiatowy w Chmielniku, Chmielknik, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61afb7c6f571d4002a64b469